CLINICAL TRIAL: NCT06150235
Title: Impact of Physical Activity on Quality of Life for Chronic Hemodialysis Patients
Acronym: QDV-HD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_010_QDV-HD
Record Dates: First submitted 2023-11-20; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Hemodialysis
Keywords: Quality of life; chronic hemodialysis patients; factors associated; physical activity
MeSH Terms: conditions — Motor Activity | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic hemodialysis patients: patients with chronic hemodialysis
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection

SUMMARY:
Chronic end-stage renal disease has a significant impact on patients' quality of life. In 2005, a study evaluating the quality of life of patients with end-stage chronic kidney disease using the SF-36 and KDQoL questionnaires showed that the proportion of patients with an altered quality of life varied from 20% to 50% in the physical component dimensions and from 12% to 47% in the mental component dimensions. More than 75% of dialysis patients had at least one of the 8 scores below the threshold that defines impaired quality of life. In 2011, the Quavi-REIN study involved 1251 dialysis patients showed a significant reduction of quality of life assessed using the generic SF36 questionnaire compared with the general population, in the physical and mental dimensions.

Moreover, in France, more than one senior citizens aged between 55 and 74 in three does not comply with the World Health Organisation's recommendations on the minimum level of physical activity required per day. A sedentary lifestyle is a major public health problem. It is the 4thrisk factor for mortality after hypertension, smoking and diabetes. This inactivity increases mortality and morbidity rates in humans, and consequently the risk of diseases such as cancer and type 2 diabetes.

Physical activity is recommended for patients with chronic kidney disease. In a survey of 505 nephrologists, 97% thought that physical activity is beneficial for dialysis patients, given that a sedentary lifestyle increases the death rate among dialysis patients. Data from the international DOPPS registry, involving 20,920 patients, showed that patients who engage in physical activity have a better quality of life (physical, psychological and sleep quality components), as assessed by the KDQoL-SF questionnaire.

DETAILED DESCRIPTION:
The main objective is to study factors associated with the quality of life of hemodialysis patients, including physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis
* Major
* Agreeing to participate in the study

Exclusion Criteria:

* On peritoneal dialysis
* On daily dialysis at home
* Minors
* Protected by law (guardianship, curatorship, safeguarding of justice)
* Refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life using SF-36 survey | Day 0
  Health-related quality of life will be evaluated by the generic questionnaire "Medical Outcomes Study ShortForm General Health Survey" (SF-36) created in 1992 by Ware and Sherbourne and validated in French by Leplège in 1998 The SF-36 is a questionnaire containing 36 items, covering the four weeks preceding the time when the subject is interviewed, grouped into 8 dimensions.
  Each question is assessed on a Likert scale, with 3, 5 or 6 possible answer levels.
  The score for each dimension varies from 0 to 100, the higher the score and the better the quality of life.

SECONDARY OUTCOMES:
Health-related quality of life using KDQOL survey | Day 0
  It will be evaluated by the questionnaire to chronic kidney disease proposed to patients will be the KDQOL. It will be used in its simplified version of 24 items, divided into 3 dimensions:
  symptoms and health problems: 12 items; effects of kidney disease: 8 items; burden of kidney disease: 4 items Each question has 5 to 6 possible answer levels, with ratings on a Likert scale ranging from 1 to 5 (excellent/bad) or 1 to 6 (all the time/never). A score is calculated for each dimension and corresponds to the sum of the scores of the questions constituting the dimension, divided by the number of questions for that dimension (average of the scores of the questions). If the answer to a question is missing, it is not taken into account in the calculation of the dimension score.The score for each dimension varies from 0 to 100, the higher the score and the better the quality of life.
Physical activity using RICCI GAGNON test | Day 0
  Physical activity will be evaluated by the RICCI GAGNON test .
  The RICCI GAGNON test is a questionnaire containing 9 questions. Each question is coded from 1 to 5 giving a score out of 45 points. Interpretation is as follows: under 18: inactive; between 18 and 35: active; over 35: very active.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided